CLINICAL TRIAL: NCT01057940
Title: A Pilot Study to Assess the Feasibility of Double Balloon Enteroscopy as a Rescue Technique for Failed Direct Percutaneous Endoscopic Jejunostomy Tube Placement
Brief Title: Pilot to Assess DBE as a Rescue Technique for Failed PEJ
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Louis-Michel Wong Kee Song, MD, Mayo Clinic
Other Study IDs: 09-008410
Record Dates: First submitted 2010-01-27; First posted 2010-01-28 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2013-06

CONDITIONS: Patients Who Have Failed Conventional DPEJ Placement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PEJ placement: Patients who have failed conventional DPEJ placement and would otherwise require surgical intervention.
  Interventions: Procedure: DBE PEJ placement

INTERVENTIONS:
Procedure: DBE PEJ placement — One time procedure with follow-up telephone call.

SUMMARY:
Is DBE(double balloon enteroscopy)-assisted DPEJ(direct percutaneous endoscopic jejunostomy) a viable option in patients who have failed conventional DPEJ placement and who otherwise would require surgical jejunostomy or parenteral nutrition.

DETAILED DESCRIPTION:
DBE-assisted DPEJ is a viable option in patients who have failed conventional DPEJ placement and who otherwise would require surgical jejunostomy or parenteral nutrition.

ELIGIBILITY:
Patients:

Patients who have failed conventional DPEJ tube placement will be offered participation in the study. DBE-assisted DPEJ will be performed on a subsequent day following failed DPEJ. Patients who do not wish to undergo an attempt at DBE-assisted DPEJ will follow-up with their primary caregiver for alternative means of feeding tube placement (e.g., surgical jejunostomy).

Inclusion criteria:

1. Age > 18 years old
2. Appropriate indication for DPEJ tube placement and Nutrition consult approval
3. Absence of bleeding disorder
4. Platelet count > 50,000 and INR < 1.5
5. Ability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have failed conventional DPEJ placement
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-04; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Louis Wong kee song, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States